CLINICAL TRIAL: NCT06483854
Title: Know Your Status: A Cluster Randomized Controlled Trial Comparing Healer-initiated HIV Counseling and Testing to Standard of Care in Rural South Africa
Brief Title: Healer-initiated HIV Counseling and Testing Versus Standard of Care in Rural South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Carolyn Audet, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R01MH135738 (NIH)
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hiv
Keywords: HIV counseling and testing; traditional healer practitioners
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): people who receive HIV testing in this arm through standard programs provided by clinics.
- Healer-provided (Experimental): Traditional healers will provide HIV counseling and testing services to their clients
  Interventions: Diagnostic Test: HIV counseling and testing from a traditional health practitioner

INTERVENTIONS:
Diagnostic Test: HIV counseling and testing from a traditional health practitioner — Healer provided HIV counseling and testing services offered to clients
  Arms: Healer-provided

SUMMARY:
South Africa has made progress towards their 95-95-95 goals, yet a substantial proportion of the population do not test regularly. To reach people who otherwise may avoid testing, we propose to build on our successful healer-initiated HIV counseling and testing pilot to conduct a cluster randomized controlled trial in 42 clinical catchment areas to evaluate an expanded Healer-Initiated HIV Testing and Linkage to Care intervention in rural South Africa.

DETAILED DESCRIPTION:
South Africa has made progress towards their 95-95-95 goals, yet a substantial proportion of the population do not test regularly. In South Africa, people of low socioeconomic status, men, people in rural areas, and those who distrust the health system have higher rates of HIV stigma and are less likely to receive an HIV test. These individuals are also more likely to see a traditional healer for their health care needs, making healers an ideal group to bridge the health care utilization divide.

To reach people who otherwise may avoid testing, the team trained 15 traditional healers to conduct HIV counseling and testing in their own "clinics"- a hut or room by their home where they provide care to their patients (R34MH122259-01). Over six-months, with no advertisement or community events, healers offered HIV counseling and testing to 463 individuals who visited them for unrelated services. Fifty-four (11.7%) self-reported a positive HIV status. Of the 409 eligible participants, 316 (77%) agreed to test, and 20 (6.3%) tested positive- 95% were linked to HIV care and treatment services.

In collaboration with the Department of Health and the healer's organization, this study will build on a successful pilot to test an expanded Healer-Initiated HIV Testing and Linkage to Care intervention with the following testing and linkage to care components. Healers will provide three testing services: (1) Advertise the availability of free healer-initiated counseling and testing for their clients; (2) Offer partner-based testing services at their facilities or client homes; and (3) Provide monthly community-based testing outreach activities at local events (e.g., sporting events, fairs). In addition to testing, healers will support linkage to care and treatment adherence, offering clients accompaniment to their first clinical appointment, ongoing adherence support/counseling in person or via WhatsApp, and a nurse/community health worker/healer WhatsApp group to facilitate more technical support if needed. This is a cluster randomized controlled trial (comparing standard of care (SOC) testing options vs. SOC + enhanced testing with support of traditional healers) at 42 clinical catchment areas to evaluate the impact this intervention.

The Specific Aims of this study are to: (1) Compare rates of HIV testing in healer-initiated HIV counseling and testing communities vs. control communities via a cluster randomized controlled trial in rural South Africa; (2) Assess adoption, implementation fidelity and maintenance of healer-initiated HIV testing; and (3) Evaluate the cost-effectiveness of healer-initiated HIV counseling and testing compared to standard of care. This team has a proven record of engaging traditional healers to improve patient outcomes, conducting research to evaluate and address mistrust in the health system, HIV stigma, and developing interventions to increase HIV testing uptake. Traditional healers are an untapped resource with the potential to reach those who historically avoid HIV testing and they have the potential to help South Africa reach their 95% testing targets.

ELIGIBILITY:
Inclusion Criteria:

* Community members > 18 years of age, who chose to receive an HIV test from a traditional healer.

Exclusion Criteria:

* Community members who are not of sound mind or body during the recruitment (inebriated, experiencing a mental health issue).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230907 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of HIV counseling and testing | 24 months
  At the time of a healer visit, we will assess the % of people who receive an HIV test divided by the total number of people who are invited to test and who are eligible.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Audet, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Bushbuckridge, Agincourt, MP, South Africa

IPD SHARING:
Plan to Share IPD: No